CLINICAL TRIAL: NCT04616313
Title: Novel Pulmonary Imaging of Lung Structure and Function in Symptomatic and Asymptomatic E-cigarette Smokers
Brief Title: Novel Pulmonary Imaging of Lung Structure and Function in E-cigarette Smokers
Status: Recruiting | Type: Observational
Sponsor: Western University, Canada (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Grace Parraga, PhD, Scientist. Robarts Research Institute, Western University, Canada
Other Study IDs: ROB0048
Record Dates: First submitted 2020-11-02; First posted 2020-11-04 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: E Cigarette Use
Keywords: e-cigarette smoking; pulmonary function; Xenon-129; Magnetic Resonance Imaging
MeSH Terms: conditions — Vaping | interventions — Tomography, X-Ray Computed; Respiratory Function Tests; Exercise Test; Hematologic Tests; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- c-cigarette never users: Includes 70 participants who are e-cigarette users who have never smoked combustible cigarettes.
  Interventions: Diagnostic Test: Hyperpolarized Xenon-129 MRI of the lungs; Diagnostic Test: Computed Tomography (CT); Diagnostic Test: Pulmonary Function Tests (PFT); Diagnostic Test: Cardiopulmonary exercise testing (CPET); Diagnostic Test: Sputum analysis; Diagnostic Test: Blood analysis; Other: Questionnaires
- former or current c-cigarette users: Includes 70 participants who are e-cigarette users who are also former or current combustible cigarette smokers.
  Interventions: Diagnostic Test: Hyperpolarized Xenon-129 MRI of the lungs; Diagnostic Test: Computed Tomography (CT); Diagnostic Test: Pulmonary Function Tests (PFT); Diagnostic Test: Cardiopulmonary exercise testing (CPET); Diagnostic Test: Sputum analysis; Diagnostic Test: Blood analysis; Other: Questionnaires
- never smokers: Includes 10 participants who have never smoked e-cigarettes or combustible cigarettes.
  Interventions: Diagnostic Test: Hyperpolarized Xenon-129 MRI of the lungs; Diagnostic Test: Computed Tomography (CT); Diagnostic Test: Pulmonary Function Tests (PFT); Diagnostic Test: Cardiopulmonary exercise testing (CPET); Diagnostic Test: Sputum analysis; Diagnostic Test: Blood analysis; Other: Questionnaires

INTERVENTIONS:
Diagnostic Test: Hyperpolarized Xenon-129 MRI of the lungs — Participants will be imaged using MRI using hyperpolarized xenon-129 gas as a contrast gas
  Other Names: 129Xe MRI
Diagnostic Test: Computed Tomography (CT) — Participants will undergo a CT scan of the thoracic cavity
  Other Names: CT
Diagnostic Test: Pulmonary Function Tests (PFT) — Participants will have their lung function evaluated using PFT
  Other Names: PFT
Diagnostic Test: Cardiopulmonary exercise testing (CPET) — Participants will perform cardiopulmonary exercise testing as a measure of exercise capacity
  Other Names: CPET
Diagnostic Test: Sputum analysis — Participants will provide a sputum sample that will be analysed for eosinophils
Diagnostic Test: Blood analysis — Participants will have their blood drawn and analysed for eosinophil count.
Other: Questionnaires — Participants will complete questionnaires to assess activity related dyspnea, respiratory symptoms and health status impairment and respiratory related quality of life.

SUMMARY:
This is a longitudinal study of the long-term health impact of e-cigarette smoking on the lungs. Participants will be followed over a period of 5 years, and impacts of e-cigarette smoking on the lungs will be measured with magnetic resonance imaging (MRI) using hyperpolarized xenon-129 gas, pulmonary function tests, exercise capacity, computed tomography images and questionnaires.

DETAILED DESCRIPTION:
This is a 5-year longitudinal study of the long-term lung health impact of e-cigarette smoking. Participants with a history of e-cigarette smoking age ≥ 16 years will be recruited from within 2 hours of London, ON through local family and tertiary care physicians, emergency departments and community and social media advertisements. Asymptomatic age and sex-matched participants who have never smoked e- or c-cigarettes will be recruited through community advertisement, media and social media. Participants must satisfy all inclusion and exclusion criteria in order to participate in the study. We will compare lung health of participants at baseline, 12 weeks, 24 weeks and 48 weeks, 3 years, 4 years and 5 years with an asymptomatic control group with no history of e-cigarette or c-cigarette use. The study will involve 6 in-person visits and 1 telephone call for a health update. All measurements will be made with at least 4 hours after the last cigarette and/or vape to provide a way to practically focus on chronic and not acute effects. Pulmonary function and imaging measurements will be made before and after bronchodilator administration.

At Visit 1, informed consent will be obtained before any study related assessments or procedures are performed. Eligibility criteria will be reviewed. Safety assessments including vital signs, pulmonary function testing, hematology, sputum sampling, exercise testing, and respiratory questionnaires will be completed.

Visit 2 will take place 12 weeks after visit 1 and will include vital signs, pre and post bronchodilator pulmonary function testing, pre and post bronchodilator MRI imaging, chest CT scan, exercise testing, and questionnaires.

Visit 3 will take place at 24 weeks and will involve a telephone call to update health information as well as questionnaires.

Visit 4 will take place at 48 weeks and will involve vital signs, pre and post bronchodilator pulmonary function testing, pre and post bronchodilator MRI imaging, hematology, blood chemistry, sputum analysis, exercise testing, and questionnaires.

Visit 5 will take place at year 3 and will involve vital signs, pre and post bronchodilator pulmonary function testing, pre and post bronchodilator MRI imaging, blood draw, sputum induction and analysis, exercise testing and questionnaires.

Visit 6 will take place at year 4 and will involve vital signs, pre and post bronchodilator pulmonary function testing, pre and post bronchodilator MRI imaging, blood draw, sputum induction and analysis, exercise testing and questionnaires.

Visit 7 will take place at year 5 and will involve vital signs, pre and post bronchodilator pulmonary function testing, pre and post bronchodilator MRI imaging, blood draw, sputum induction and analysis, exercise testing and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be directly obtained from legally competent participants before any study-related assessment is performed.
* Male and female participant age ≥16 years.
* Participant has recently started vaping, >1 and <5 years weekly use.
* 70 participants will be c-cigarette never users.
* 70 participants will be former or current c-cigarette users.
* 10 asymptomatic age and sex-matched healthy people who have never used e- or c-cigarettes will be controls.

Exclusion Criteria:

* Participants with contraindications for undergoing an MRI such as participants with MRI-sensitive implants, tattoos with MRI-sensitive dye and severe claustrophobia.
* Participant is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand written material.
* Participant unable to perform spirometry or plethysmography maneuvers.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. e-cigarette users who did not require hospitalization, nor used c-cigarettes
  2. e-cigarette users who also consumed c-cigarettes
  3. never smokers
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Determine if e-cigarette users who did not require hospitalization, nor used c-cigarettes report pulmonary imaging abnormalities. | 12 weeks following enrollment
  Measured using 129-Xe MRI
Determine if e-cigarette users who did not require hospitalization, nor used c-cigarettes report pulmonary imaging abnormalities. | 12 weeks following enrollment
  Measured using computed tomography imaging
Determine if e-cigarette users who did not require hospitalization, nor used c-cigarettes report respiratory symptoms or abnormal pulmonary function measured by FEV1. | 12 weeks following enrollment
  Measured using forced expiratory volume in one second (FEV1)
Determine if e-cigarette users who did not require hospitalization, nor used c-cigarettes report respiratory symptoms or abnormal pulmonary function measured by FVC. | 12 weeks following enrollment
  Measured using forced vital capacity (FVC)
Determine if e-cigarette users who did not require hospitalization, nor used c-cigarettes report respiratory symptoms or abnormal pulmonary function measured by TLC. | 12 weeks following enrollment
  Measured using total lung capacity (TLC)
Determine if e-cigarette users who did not require hospitalization, nor used c-cigarettes report respiratory symptoms or abnormal pulmonary function measured by FRC. | 12 weeks following enrollment
  Measured using functional residual capacity (FRC)
Determine if e-cigarette users who did not require hospitalization, nor used c-cigarettes report respiratory symptoms or abnormal pulmonary function measured by RV. | 12 weeks following enrollment
  Measured using residual volume (RV)
Determine if e-cigarette users who did not require hospitalization, nor used c-cigarettes report respiratory symptoms or abnormal pulmonary function measured by FOT. | 12 weeks following enrollment
  Measured using forced oscillation technique (FOT)
Determine if e-cigarette users who did not require hospitalization, nor used c-cigarettes report respiratory symptoms or abnormal pulmonary function measured by LCI. | 12 weeks following enrollment
  Measured using lung clearance index (LCI)
Determine if e-cigarette users who did not require hospitalization, nor used c-cigarettes report respiratory symptoms or abnormal pulmonary function measured by FeNO. | 12 weeks following enrollment
  Measured using Fractional Exhaled Nitric Oxide (FeNO).
Determine if e-cigarette users who did not require hospitalization, nor used c-cigarettes report respiratory symptoms or abnormal pulmonary function measured by exercise capacity | 12 weeks following enrollment
  Exercise capacity measured by cardio-pulmonary exercise testing (CPET)

SECONDARY OUTCOMES:
Differences in airways between e-cigarette-only smokers and both e-cigarette and c-cigarette smokers. | 5 years
  Measured using 129-Xe MRI
Differences in airways between e-cigarette-only smokers and never smokers. | 5 years
  Measured using 129-Xe MRI
Differences in parenchyma between e-cigarette-only smokers and both e-cigarette and c-cigarette smokers. | 5 years
  Measured using 129-Xe MRI
Differences in parenchyma between e-cigarette-only smokers and never smokers. | 5 years
  Measured using 129-Xe MRI
Changes in airways of e-cigarette smokers over time. | 5 years
  Measured using Xenon-129 (129-Xe) MRI
Changes in parenchyma of e-cigarette smokers over time. | 5 years
  Measured using Xenon-129 (129-Xe) MRI
Changes in lung function of e-cigarette smokers over time as measured by FEV1. | 5 years
  Measured using forced expiratory volume in one second (FEV1).
Changes in lung function of e-cigarette smokers over time as measured by FVC. | 5 years
  Measured using forced vital capacity (FVC)
Changes in lung function of e-cigarette smokers over time as measured by TLC. | 5 years
  Measured using total lung capacity (TLC)
Changes in lung function of e-cigarette smokers over time as measured by FRC. | 5 years
  Measured using functional residual capacity (FRC)
Changes in lung function of e-cigarette smokers over time as measured by RV. | 5 years
  Measured using residual volume (RV)
Changes in lung function of e-cigarette smokers over time as measured by FOT. | 5 years
  Measured using forced oscillation technique (FOT).
Changes in lung function of e-cigarette smokers over time as measured by LCI. | 5 years
  Measured using lung clearance index (LCI)
Changes in lung function of e-cigarette smokers over time as measured by FeNO. | 5 years
  Measured using Fractional Exhaled Nitric Oxide (FeNO)
Changes in lung function of e-cigarette smokers over time as measured by exercise capacity. | 5 years
  Exercise capacity measured by cardio-pulmonary exercise testing (CPET)
Changes in lung health of e-cigarette smokers over time as measured by the mMRC dyspnea scale questionnaire. | 5 years
  Measured using the modified medical research council (mMRC) dyspnea scale
Changes in lung health of e-cigarette smokers over time as measured by SGRQ. | 5 years
  Measured using the St. George's respiratory questionnaire (SGRQ)
Changes in lung health of e-cigarette smokers over time as measured by CAT. | 5 years
  Measured using the COPD assessment test (CAT)
Changes in lung health of e-cigarette smokers over time as measured by IPAQ. | 5 years
  Measured using the International Physical Activity Questionnaire (IPAQ).

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, Principal Investigator — Western University - Robarts Research Institute
Locations (1):
- Robarts Research Institute; The University of Western Ontario; London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hua M, Alfi M, Talbot P. Health-related effects reported by electronic cigarette users in online forums. J Med Internet Res. 2013 Apr 8;15(4):e59. doi: 10.2196/jmir.2324. PMID 23567935
- [Background] Wang MP, Ho SY, Leung LT, Lam TH. Electronic Cigarette Use and Respiratory Symptoms in Chinese Adolescents in Hong Kong. JAMA Pediatr. 2016 Jan;170(1):89-91. doi: 10.1001/jamapediatrics.2015.3024. No abstract available. PMID 26551991
- [Background] McConnell R, Barrington-Trimis JL, Wang K, Urman R, Hong H, Unger J, Samet J, Leventhal A, Berhane K. Electronic Cigarette Use and Respiratory Symptoms in Adolescents. Am J Respir Crit Care Med. 2017 Apr 15;195(8):1043-1049. doi: 10.1164/rccm.201604-0804OC. PMID 27806211
- [Background] Cho JH, Paik SY. Association between Electronic Cigarette Use and Asthma among High School Students in South Korea. PLoS One. 2016 Mar 4;11(3):e0151022. doi: 10.1371/journal.pone.0151022. eCollection 2016. PMID 26942764
- [Background] Schweitzer RJ, Wills TA, Tam E, Pagano I, Choi K. E-cigarette use and asthma in a multiethnic sample of adolescents. Prev Med. 2017 Dec;105:226-231. doi: 10.1016/j.ypmed.2017.09.023. Epub 2017 Sep 28. PMID 28964850
- [Background] Layden JE, Ghinai I, Pray I, Kimball A, Layer M, Tenforde MW, Navon L, Hoots B, Salvatore PP, Elderbrook M, Haupt T, Kanne J, Patel MT, Saathoff-Huber L, King BA, Schier JG, Mikosz CA, Meiman J. Pulmonary Illness Related to E-Cigarette Use in Illinois and Wisconsin - Final Report. N Engl J Med. 2020 Mar 5;382(10):903-916. doi: 10.1056/NEJMoa1911614. Epub 2019 Sep 6. PMID 31491072
- [Background] Henry TS, Kanne JP, Kligerman SJ. Imaging of Vaping-Associated Lung Disease. N Engl J Med. 2019 Oct 10;381(15):1486-1487. doi: 10.1056/NEJMc1911995. Epub 2019 Sep 6. No abstract available. PMID 31491070
- [Background] Maddock SD, Cirulis MM, Callahan SJ, Keenan LM, Pirozzi CS, Raman SM, Aberegg SK. Pulmonary Lipid-Laden Macrophages and Vaping. N Engl J Med. 2019 Oct 10;381(15):1488-1489. doi: 10.1056/NEJMc1912038. Epub 2019 Sep 6. No abstract available. PMID 31491073
- [Background] Davidson K, Brancato A, Heetderks P, Mansour W, Matheis E, Nario M, Rajagopalan S, Underhill B, Wininger J, Fox D. Outbreak of Electronic-Cigarette-Associated Acute Lipoid Pneumonia - North Carolina, July-August 2019. MMWR Morb Mortal Wkly Rep. 2019 Sep 13;68(36):784-786. doi: 10.15585/mmwr.mm6836e1. PMID 31513559
- [Background] Landman ST, Dhaliwal I, Mackenzie CA, Martinu T, Steel A, Bosma KJ. Life-threatening bronchiolitis related to electronic cigarette use in a Canadian youth. CMAJ. 2019 Dec 2;191(48):E1321-E1331. doi: 10.1503/cmaj.191402. Epub 2019 Nov 20. PMID 31753841
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Oostveen E, MacLeod D, Lorino H, Farre R, Hantos Z, Desager K, Marchal F; ERS Task Force on Respiratory Impedance Measurements. The forced oscillation technique in clinical practice: methodology, recommendations and future developments. Eur Respir J. 2003 Dec;22(6):1026-41. doi: 10.1183/09031936.03.00089403. PMID 14680096
- [Background] Kirby M, Heydarian M, Svenningsen S, Wheatley A, McCormack DG, Etemad-Rezai R, Parraga G. Hyperpolarized 3He magnetic resonance functional imaging semiautomated segmentation. Acad Radiol. 2012 Feb;19(2):141-52. doi: 10.1016/j.acra.2011.10.007. Epub 2011 Nov 21. PMID 22104288
- [Background] Owrangi AM, Etemad-Rezai R, McCormack DG, Cunningham IA, Parraga G. Computed tomography density histogram analysis to evaluate pulmonary emphysema in ex-smokers. Acad Radiol. 2013 May;20(5):537-45. doi: 10.1016/j.acra.2012.11.010. PMID 23570935
- [Background] Pizzichini E, Pizzichini MM, Efthimiadis A, Evans S, Morris MM, Squillace D, Gleich GJ, Dolovich J, Hargreave FE. Indices of airway inflammation in induced sputum: reproducibility and validity of cell and fluid-phase measurements. Am J Respir Crit Care Med. 1996 Aug;154(2 Pt 1):308-17. doi: 10.1164/ajrccm.154.2.8756799.
- [Background] McGavin CR, Artvinli M, Naoe H, McHardy GJ. Dyspnoea, disability, and distance walked: comparison of estimates of exercise performance in respiratory disease. Br Med J. 1978 Jul 22;2(6132):241-3. doi: 10.1136/bmj.2.6132.241. PMID 678885
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Jones PW, Quirk FH, Baveystock CM, Littlejohns P. A self-complete measure of health status for chronic airflow limitation. The St. George's Respiratory Questionnaire. Am Rev Respir Dis. 1992 Jun;145(6):1321-7. doi: 10.1164/ajrccm/145.6.1321. PMID 1595997
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694